CLINICAL TRIAL: NCT00349297
Title: The Microbiological Spectrum in Acute Dacryocystitis
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Other Study IDs: R325/18/2003
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Dacryocystitis
MeSH Terms: conditions — Dacryocystitis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Acute dacryocystitis in adults can be a very painful disease and may not respond well to medical therapy.

The purpose of this prospective non-randomised study is to determine the microorganisms causing acute dacryocystitis and the antibiotic sensitivities of these organisms.

The study also aims to correlate the microbiological findings to the severity of clinical manifestations and evaluate the effectiveness of our current practice of aspiration and empiric systemic antibiotic therapy in treating patients with acute dacryocystitis and hence review whether there is a need to alter current management strategy.

ELIGIBILITY:
INCLUSION CRITERIA:

* Painful localised fluctuant induration just inferior to the medial canthal tendon of less than 2 weeks duration.

EXCLUSION CRITERIA:

* Non-fluctuant lacrimal sac swelling
* Uncooperative patient
* Unwilling Patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute dacryocystitis patients
Sampling Method: Non-Probability Sample
Dates: Start 2003-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anshu Arundhati, MRCSED, MMED, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore